CLINICAL TRIAL: NCT03427060
Title: CONSENT II: Coversin in Paroxysmal Nocturnal Hemoglobinuria (PNH) in Patients With Resistance to Eculizumab Due to Complement C5 Polymorphisms
Brief Title: Coversin in PNH in Patients With Resistance to Eculizumab Due to Complement C5 Polymorphisms
Acronym: CONSENTII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AKARI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK585
Record Dates: First submitted 2018-01-24; First posted 2018-02-09 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Coversin treatment (Experimental): Coversin - 22.5mg followed by 45mg for 6 months.
  Interventions: Drug: Coversin

INTERVENTIONS:
Drug: Coversin — Coversin - 22.5mg followed by 45mg for 6 months.

SUMMARY:
Coversin in Paroxysmal Nocturnal Hemoglobinuria (PNH) in patients with resistance to Eculizumab due to complement C5 polymorphisms.

DETAILED DESCRIPTION:
Coversin, a small protein complement C5 inhibitor which prevents the cleavage of C5 by C5 convertase into C5a and C5b, will be used in an open label, non-comparative clinical trial in patients with PNH and proven resistance to eculizumab due to C5 polymorphisms. Patients will be treated with Coversin by daily subcutaneous injection for 6 months in order to determine the safety and efficacy of the drug in these circumstances. If satisfactory control of the PNH is achieved, and at the discretion of the Principal Investigator (PI), patients will have the option of remaining on Coversin and being entered into the long term follow-up study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with known PNH.
2. Aged 18 and above. No upper age limit.
3. Lactate dehydrogenase (LDH) ≥1.5 upper limit of normal.
4. Must agree to use two methods of contraception that are ≥99% effective in preventing pregnancy.
5. Resistance to eculizumab (Soliris®).
6. Voluntary written informed consent.
7. Willing to self-inject Coversin daily.
8. Willing to receive appropriate prophylaxis against Neisseria infection.
9. Willing to avoid prohibited medications for duration of study.

Exclusion Criteria:

1. Subjects with body weight <50 kg (110 lb) or >100 kg (220 lb).
2. Pregnancy or breast feeding (females).
3. Known allergy to ticks or severe reaction to arthropod venom (e.g. bee or wasp venom).
4. Unresolved Neisseria meningitidis infection.
5. Patients who have not received adequate immunization against Neisseria meningitides.
6. Impaired hepatic function.
7. Patients with impaired renal function.
8. Failure to satisfy the Principal Investigator (PI) of fitness to participate for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2021-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with paroxysmal nocturnal hemoglobinuria (PNH) who had received eculizumab without apparent benefit and in whom it had been demonstrated that their serum was resistant to eculizumab at any concentration (due to complement C5 polymorphisms that prevent tight binding of eculizumab) were recruited from one medical center between May 2018 and February 2021.
Pre-assignment Details: There were no patients excluded from the study following enrolment
Groups:
- Coversin Treatment: This is an open label, non-comparator study.
  Patients were to receive coversin at ablation, initiation and maintenance doses:
  * Ablation (Day 1): 60 mg and 30 mg (12 hours apart)
  * Initiation (Day 2 - 28): 22.5 mg twice a day
  * Maintenance (Day 29 - 180): 45 mg once daily
Period: Overall Study
Arm/Group | Coversin Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Coversin Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Height [Number; unit: cm] | 155
Weight [Number; unit: kg] | 73.3

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Serum Lactate Dehydrogenase (LDH)
Description: Measurement of serum lactate dehydrogenase (LDH)
Time Frame: Baseline to Day 186
Measure: Number; unit: U/L
Arm/Group | Coversin Treatment
Number analyzed (Participants) | 1
U/L
  Screening | 2913
  Day 1 | 3056
  Day 3 | 1453
  Day 7 | 564
  Day 14 | 351
  Day 21 | 368
  Day 29 | 329
  Day 36 | 339
  Day 43 | 555
  Day 60 | 319
  Day 90 | 394
  Day 120 | 352
  Day 150 | 284
  Day 183 | 906
  Day 184 | 882
  Day 186 | 612

2. Secondary Outcome: Percentage Change in Haemoglobin (Hb) Compared to Screening
Description: Percentage change in the haemoglobin (Hb) value at each study visit compared to screening
Time Frame: Baseline to Day 186
Measure: Number; unit: %change in Hb value compare to screening
Arm/Group | Coversin Treatment
Number analyzed (Participants) | 1
%change in Hb value compare to screening
  Screening | 0
  Day 1 | 28
  Day 3 | 18
  Day 7 | 22
  Day 14 | 17
  Day 21 | 25
  Day 29 | 23
  Day 36 | 9
  Day 43 | 26
  Day 60 | 60
  Day 90 | 28
  Day 120 | 18
  Day 150 | 23
  Day 186 | 26

3. Secondary Outcome: Number of Packed Red Blood Cells (PRBC) Transfusions
Description: Number of units of packed red blood cells (PRBC) transfusions
Time Frame: Baseline to Day 180
Measure: Number; unit: PRBC Units
Arm/Group | Coversin Treatment
Number analyzed (Participants) | 1
PRBC Units
  Day -35 | 1
  Day -10 | 2
  Day 38 | 1
  Day 39 | 2

ADVERSE EVENTS:
Time Frame: All adverse events were collected from the time of informed consent until completion of patient's study participation. From Screening to Day 186
Groups:
- Coversin Treatment. Ablation Dose: Day 1. 60 mg and 30 mg (12 Hours Apart); Coversin Treatment. Initiation Dose: Days 2 - 28. 22.5 mg Twice a Day (12 Hours Apart); Coversin Treatment. Maintenance Dose: Days 29 - 180. 45 mg Once Daily: This is an open label, non-comparator study.
  Patients were to receive coversin at ablation, initiation and maintenance doses:
  * Ablation (Day 1): 60 mg and 30 mg (12 hours apart)
  * Initiation (Day 2 - 28): 22.5 mg twice a day
  * Maintenance (Day 29 - 180): 45 mg once daily
Arm/Group | Coversin Treatment. Ablation Dose: Day 1. 60 mg and 30 mg (12 Hours Apart) | Coversin Treatment. Initiation Dose: Days 2 - 28. 22.5 mg Twice a Day (12 Hours Apart) | Coversin Treatment. Maintenance Dose: Days 29 - 180. 45 mg Once Daily
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coversin Treatment. Ablation Dose: Day 1. 60 mg and 30 mg (12 Hours Apart) (N=1) | Coversin Treatment. Initiation Dose: Days 2 - 28. 22.5 mg Twice a Day (12 Hours Apart) (N=1) | Coversin Treatment. Maintenance Dose: Days 29 - 180. 45 mg Once Daily (N=1)
Device related Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Catheter-related infection
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coversin Treatment. Ablation Dose: Day 1. 60 mg and 30 mg (12 Hours Apart) (N=1) | Coversin Treatment. Initiation Dose: Days 2 - 28. 22.5 mg Twice a Day (12 Hours Apart) (N=1) | Coversin Treatment. Maintenance Dose: Days 29 - 180. 45 mg Once Daily (N=1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT03427060/Prot_SAP_000.pdf